CLINICAL TRIAL: NCT03566459
Title: Making Medication Assisted Treatment Available to Veterans With Opioid Use Disorders at CBOCs Using Telemedicine (PII 18-178)
Brief Title: Medications for Opioid Use Disorders (MOUD) Via Telemedicine
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: PIX 18-001; PII 18-178 (Other Grant/Funding Number: QUERI)
Record Dates: First submitted 2018-04-10; First posted 2018-06-25 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder (OUD); Medication Assisted Treatment (MAT); Telemedicine; Veteran
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Veterans with opioid use disorder (OUD): Veterans with opioid use disorder (OUD) in VA Maine Healthcare System catchment area
  Interventions: Other: CBOC offering Tele-MOUD to Veterans; Other: CBOC not offering Tele-MOUD to Veterans

INTERVENTIONS:
Other: CBOC offering Tele-MOUD to Veterans — CBOC offering medications for opioid use disorder (MOUD) using telemedicine
Other: CBOC not offering Tele-MOUD to Veterans — CBOC not offering medications for opioid use disorder (MOUD) using telemedicine

SUMMARY:
Medication Assisted Treatment (MAT) of Veterans with Opioid Use Disorder (OUD) decreases mortality and improves treatment follow-up. However, outside of large and/or urban VA medical centers, there are shortages of providers with experience treating OUD and a license to prescribe buprenorphine. This has resulted in decreased access to MAT (buprenorphine/naloxone and injectable naltrexone) at rural CBOCs and increased overdose rates in rural areas. Some individual prescribers have used clinical video teleconferencing (CVT) to overcome geographic barriers and prescribe MAT to Veterans in CBOCs. However, while locally effective, these arrangements are not standardized and are not parts of larger VISN-wide or national VHA strategies.

This proposal describes an effective program that the investigators propose to replicate and expand. The program involves increasing prescribing rates of MAT for OUD in CBOCs using telemedicine. The investigators propose to (A) develop materials and procedures for the dissemination of telemedicine delivery of MAT to Veterans at CBOCs and (B) implement telemedicine prescribing of MAT at rural CBOCs in Northern Maine that lack on-site MAT providers. MAT will be prescribed by the VISN 1 Telemental Health Hub, which already provides medication management, psychotherapy, and some MAT to sites in Northern Maine.

In later years, the program will be expanded to other VISN 1 CBOCs, and to other TMH Regional Hubs that provide services to wide catchment areas in other VISNs. By building on an existing infrastructure connecting these TMH Regional Hubs to CBOCs and collaborating with other national initiatives (e.g. SCAN ECHO, PDSI, and academic detailing), telemedicine MAT will be rapidly disseminated to Veterans at CBOCs who are at high risk for illness, overdose, and premature death from opioids.

DETAILED DESCRIPTION:
Medication Assisted Treatment (MAT) of Veterans with Opioid Use Disorder (OUD) decreases mortality and improves treatment follow-up. However, outside of large and/or urban VA medical centers, there are shortages of providers with experience treating OUD and a license to prescribe buprenorphine. This has resulted in decreased access to MAT (buprenorphine/naloxone and injectable naltrexone) at rural CBOCs and increased overdose rates in rural areas. Some individual prescribers have used clinical video teleconferencing (CVT) to overcome geographic barriers and prescribe MAT to Veterans in CBOCs. However, while locally effective, these arrangements are not standardized and are not parts of larger VISN-wide or national VHA strategies.

This proposal describes an effective program that the investigators propose to replicate and expand. The program involves increasing prescribing rates of MAT for OUD in CBOCs using telemedicine. The investigators propose to (A) develop materials and procedures for the dissemination of telemedicine delivery of MAT to Veterans at CBOCs and (B) implement telemedicine prescribing of MAT at rural CBOCs in Northern Maine that lack on-site MAT providers. MAT will be prescribed by the VISN 1 Telemental Health Hub, which already provides medication management, psychotherapy, and some MAT to sites in Northern Maine.

In later years, the program will be expanded to other VISN 1 CBOCs, and to other TMH Regional Hubs that provide services to wide catchment areas in other VISNs. By building on an existing infrastructure connecting these TMH Regional Hubs to CBOCs and collaborating with other national initiatives (e.g. SCAN ECHO, PDSI, and academic detailing), telemedicine MAT will be rapidly disseminated to Veterans at CBOCs who are at high risk for illness, overdose, and premature death from opioids.

The "Replicating Existing Programs with Blended (External and Internal) Facilitation" approach will be the study's implementation strategy. Existing programs of telemedicine MAT---including those by VA Maine and VISN 1 TMH Regional Hub prescribers---will be replicated. External Facilitation, an approach that has been effective in increasing intervention uptake in controlled trials, will be provided to rural CBOCs in Northern Maine by expert study investigators. Internal Facilitation will be provided by VA Maine primary care and pharmacy staff, who are already supporting programs in opioid prescribing safety in the VA Maine Healthcare System. Supporting this project are consultants and collaborators with expertise in implementation science, program evaluation, pain treatment, academic detailing, and telemedicine MAT. Data collected during implementation will inform program expansion. The primary measure of program outcomes will be the SAIL SUD16 measure of MAT use for Veterans with OUD.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with OUD

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Veterans with OUD
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Population potentially able to benefit from telemedicine MAT | through study completion, up to 1 year
  Review Veterans with OUD at CBOC and compare those referred to telemedicine MAT to those not referred.
  Note that OUD diagnosis may increase over time with better OUD detection
AUDIT-C | through study completion, up to 1 year
  The Alcohol Use Disorders Identification Test is a ten-question test developed by a World Health Organization-sponsored collaborative project to determine if a person may be at risk for alcohol abuse problems.
Cost of Telemedicine MAT | through study completion, up to 1 year
  cost of time provider and other staff spent in service delivery preparing for and interacting with patients (prompted by CPT-coded encounters). Costs are calculated by multiplying time by personnel costs.
Cost of Training and Implementation | through study completion, up to 1 year
  cost of time spent by External and Internal facilitators on training/implementation. Time-spent will be assessed by weekly questions about a list of possible training activities.
Veterans' subjective experience of telemedicine MAT | through study completion, up to 1 year
  Interviews with treated Veterans covering the following topics (9): how came to program, other options considered; experience of intake, of induction onto MAT, of maintenance tele-prescribing visits, of other addiction treatment; good things/not-so-good things about treatment, recommended improvements, how compares to in-person treatment.
Providers' experience of implementing MAT | through study completion, up to 1 year
  Key informant interviews after implementation with hub and spoke providers, as described earlier.
Negative toxicology tests | through study completion, up to 1 year
  % toxicology tests that are negative for illicit opioids
Number of CBOCs participating in telemedicine MAT | through study completion, up to 1 year
  Number of CBOCs utilizing telemedicine MAT
Brief Addiction Monitor-Revised (BAM-R) | through study completion, up to 1 year
  Brief Addiction Monitor-Revised (BAM-R) upon intake and two months later.
Number of providers participating in telemedicine MAT | through study completion, up to 1 year
  Number at hubs and proportions tele-prescribing MAT; number at spokes seeing Veterans as part of their MAT treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marc I. Rosen, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Maine Healthcare System, Augusta, Maine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brunet N, Moore DT, Lendvai Wischik D, Mattocks KM, Rosen MI. Increasing buprenorphine access for veterans with opioid use disorder in rural clinics using telemedicine. Subst Abus. 2022;43(1):39-46. doi: 10.1080/08897077.2020.1728466. Epub 2020 Feb 20. PMID 32078492